CLINICAL TRIAL: NCT01956006
Title: Pilot Study of Slow Release Oral Milrinone in Patients With Advanced Heart Failure
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Alfred (Other)
Responsible Party: Principal Investigator, Prof David Kaye, Head, Experimental Cardiology and Heart Failure Division Baker Heart Research Institute & Cardiologist, Heart Centre, Alfred Hospital, The Alfred
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DK-MIL-2
Record Dates: First submitted 2013-09-25; First posted 2013-10-08 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Milrinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MIlrinone (Experimental): ER milrinone
  Interventions: Drug: Milrinone

INTERVENTIONS:
Drug: Milrinone — Administration of study medications, PK sampling and safety profile- add on haemodynamic invasive measurements if patient consents to.

SUMMARY:
Advanced heart failure (HF), ineffective pumping of the heart, is a common, life-threatening cardiovascular disorder, characterised by marked symptomatic limitation and frequent hospitalization. It is particularly prevalent in older individuals (up to 10% of the population) and it has become the most common cause for hospitalization in people >65yrs. As such it is also one of the leading consumers of healthcare spending. Recurrent hospitalization is frequently due in significant part to the lack of viable therapeutic options for severe HF. During hospital admission, medications through a drip to give through a vein (intravenous therapy), is required to improve heart pumping capacity (such as milrinone).They are frequently used and in many cases prolonged treatment periods of intravenous therapy are required. In a growing number of cases, there is a need to continue this treatment at home, however this is particularly costly and often complicated by intravenous line infection. As such there is an expanding need for therapeutic options in patients with advanced HF. Over 20 years ago, studies of the potential utility of a rapid release form of oral milrinone were examined, however these studies demonstrated adverse effects due to its quick release.

This study aims to determine the safety and tolerability of slow release oral milrinone in advanced HF patients with no further clinical option and to evaluate its effects on HF status.

ELIGIBILITY:
Inclusion Criteria:

* Advanced HF (current inpatients) with no further clinical options as defined by treating cardiologist.
* NYHA III-IV
* LVEF<35%
* Recurrent hospitalization (>/=3 admissions in the preceding 12 months) for HF
* On optimal tolerated medical/device therapy. Stable therapy for 48hrs.
* Age 18-85 yrs
* Provide written informed consent prior to any study procedure and agree to adhere to all protocol requirements

Exclusion Criteria:

* Hypotension (BPsys<85)
* Unstable rhythm including frequent non-sustained ventricular tachycardia or poorly controlled atrial fibrillation (ventricular rate >100).
* Severe renal impairment Cr>250umol/L or dialysis.
* Other life-threatening eg neoplastic, haematological, hepatic or pulmonary disease.
* Pregnancy or female with childbearing potential and inability to use contraception

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2018-05-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 3 months
  Number of MACE events change from basline safety profile bloods (Full Blood Count, urea and creatine, Liver function counts) Change in haemodynamic measurements ECG and Blood pressure and HR Monitoring Swan Ganz insertion for haemodynamic measurements (RA volume , RVSP, CO, PA, PAWP)

SECONDARY OUTCOMES:
NYHA Class | 3 months
  Change in Heart Failure Status

OTHER OUTCOMES:
6 minute walk test | 3 month
  Change in exercise capacity
BNP | 3 month
Number of Heart Failure Hospitalisation | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No